CLINICAL TRIAL: NCT05360979
Title: A Prospective, Single-arm Clinical Study of Envafolimab Combined With Chemotherapy and Recombinant Human Endostatin in Patients With Operable Stage II, IIIA, and IIIB (T3N2) Non-small Cell Lung Cancer
Brief Title: A Clinical Study of Immunotherapy Combined With Chemotherapy and Anti-angiogenic Therapy in Operable NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Second Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, xianling liu, Director of the oncology department of the Second Xiangya Hospital of Central South University, Second Xiangya Hospital of Central South University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSCLC-LXL002
Record Dates: First submitted 2021-12-26; First posted 2022-05-04 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — envafolimab; Endostatins; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant and adjuvant therapy (Experimental): After signing the informed consent, eligible subjects who meet the inclusion criteria will receive neoadjuvant therapy comprising envafolimab combined with platinum-containing chemotherapy and recombinant human endostatin, as well as postoperative envafolimab single-agent adjuvant therapy.
  Interventions: Drug: envafolimab

INTERVENTIONS:
Drug: envafolimab — Envafolimab: 300 mg, D1, Q3W, subcutaneously administered
  Other Names: recombinant human endostatin; chemotherapy

SUMMARY:
The objective of this prospective, single-arm, single-center clinical study is to evaluate the efficacy and safety of envafolimab combined with platinum-containing dual-drug chemotherapy and recombinant human endostatin regimens for treating patients with operable II, IIIA, and IIIB (T3N2) stage NSCLC.

DETAILED DESCRIPTION:
Patients with stage II, IIIA, and IIIB (T3N2) NSCLC that did not previously receive systemic treatment and can be treated with surgery were recruited. After signing the informed consent, eligible subjects who meet the inclusion criteria will receive neoadjuvant therapy comprising envafolimab combined with platinum-containing chemotherapy and recombinant human endostatin, as well as postoperative envafolimab single-agent adjuvant therapy.

During the preoperative neoadjuvant therapy period, 3 cycles of envafolimab (300 mg fixed-dose Q3W) with recombinant human endostatin (210 mg, CIV [continuous intravenous pump injection], 72 h, Q3W), and platinum-containing dual-drug chemotherapy (Q3W) will be performed, with a dosing cycle performed every 3 weeks. The study drug will be administered on the first day of each cycle.

All subjects will undergo preoperative imaging evaluation and surgical indication evaluation at 3-5 weeks after the third cycle of preoperative medication.

After completing the first 3 cycles of neoadjuvant therapy, all subjects persistently presenting indications for surgery will undergo radical surgery for NSCLC within 4-6 weeks according to the standards defined by the World Association for the Study of Lung Cancer. The pathological staging will be performed according to the AJCC Cancer Staging Manual (8th edition). Local pathologists will evaluate the surgical margins of all specimens removed during the operation. Tumor tissue samples collected from subjects during the research process will be submitted to the designated central laboratory for pathological remission assessment and translational research.

Postoperative envafolimab monotherapy (300 mg, Q3W) will be initiated at 4-6 weeks post-surgery and maintained for 1 year Adverse events (AE) will be monitored throughout the study period, and the severity of AEs will be assessed according to the guidelines listed in the National Cancer Institute (NCI) Commonly Used Terminology Criteria for Adverse Events (CTCAE) version 5.0 or above. Safety follow-ups will be conducted for all patients receiving treatment and those who warrant early discontinuation. All subjects will be followed up for OS until death, withdrawal of informed consent, or the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all following inclusion criteria to be eligible for study entry:

  1. The subjects fully understand the research and voluntarily sign the informed consent form (ICF);
  2. Subjects are aged between 18 to 70 years, irrespective of gender;
  3. Patients with resectable stage II, stage IIIA, and stage IIIB (T3N2) (AJCC staging 8th edition) NSCLC with no prior treatment and confirmed by histology; TNM staging can be confirmed by positron emission tomography (PET)-computed tomography (CT) or pathological biopsy;
  4. The presence of measurable lesions according to version 1.1 of the evaluation standard for the efficacy of solid tumors;
  5. Tumor tissue specimens can be submitted for pathological diagnosis, programmed death-ligand 1 (PD-L1) expression, and biomarker detection before enrollment (tumor tissues must be fresh specimens or archived samples obtained within three months before enrollment; tumor tissue specimen must be histological samples, including, but not limited to, puncture tissues obtained by thick and hollow needles, tissues obtained by bronchoscope clamps, or surgical removal samples. Puncture tissues obtained by fine needles and samples obtained by bronchial brushing are unacceptable);
  6. Eastern Cooperative Oncology Group (ECOG) score 0-1;
  7. Good organ function;
  8. Hematology: Absolute neutrophil count (ANC) ≥ 1500/μL; platelets ≥ 100000/μL; hemoglobin ≥ 9.0 g/dL or ≥ 5.6 mmol/L;
  9. Kidney: Serum creatinine ≤ 1.5× upper limit of normal (ULN) or calculated creatinine clearance rate (CrCl) ≥ 60 mL/min (using Cock-Gault formula);
  10. Liver: total bilirubin ≤ 1.5 × ULN or for subjects with total bilirubin level > 1.5 × ULN, direct bilirubin within normal limits; Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic-pyruvic transaminase [SGPT]) ≤ 2.5 × ULN;
  11. Endocrine system: Thyroid-stimulating hormone (TSH) is within normal limits. Note: If TSH is not within the normal range at baseline, and if T3 and free T4 are within the normal range, then the subject can be considered to meet inclusion criteria; Coagulation function: international normalized ratio (INR) or prothrombin time (PT), activation partial thromboplastin time (aPTT) ≤ 1.5 × ULN, except for cases: subjects who are receiving anticoagulant therapy, if the PT or aPTT is within the intended use range of anticoagulant drugs;
  12. Patients are willing and able to comply with the research plan's visits, treatment plans, laboratory examinations, and other research procedures;
  13. According to the assessment of the surgeon, the total lung function can withstand the planned lung resection;
  14. Women of childbearing age must undergo a serum pregnancy test within 3 days before the first treatment, and the result should be negative. Female subjects of childbearing age and male subjects whose partners are women of childbearing age must agree to use high-efficiency methods of contraception during the study and within 180 days after the last administration of the study drug.

Exclusion Criteria:

- 1. Presence of unresectable or metastatic disease; 2. Subjects with NSCLC, large cell neuroendocrine carcinoma (LCNEC), sarcomatoid tumors involving the upper sulcus; subjects with non-squamous NSCLC with known EGFR (epidermal growth factor receptor) mutations or ALK translocations; 3. Subjects with early-stage NSCLC who previously received systemic anticancer treatment, including experimental drug treatment; subjects with a history of (non-infectious) pneumonia/interstitial lung disease that requires steroid treatment, or currently present pneumonia/interstitial disease that requires steroid treatment pulmonary disease; 4. Subjects with a history of active tuberculosis; 5. Subjects with active infections requiring systemic treatment; 6. Subjects with known or suspected autoimmune diseases or immunodeficiency, except for patients with a history of hypothyroidism who do not need hormone therapy or are receiving physiological dose hormone replacement therapy; subjects with stable type I diabetes with controlled blood sugar levels; 7. Subjects with uncontrolled active hepatitis B (defined as a positive test result for hepatitis B virus surface antigen [HBsAg] during the screening period, and the detection value of HBV-DNA exceeds the ULN value of the laboratory department of the research center); (Subjects whose HBV-DNA content <500 IU/mL tested within 28 days before enrollment, and have received at least 14 days of local standard antiviral therapy and are willing to continue to receive antiviral therapy during the study period can be included); Subjects with active hepatitis C (defined as a positive test result of hepatitis C virus surface antibody [HCsAb] and HCV-RNA positive during the screening period); 8. Known human immunodeficiency virus (HIV) infection (known HIV antibody positive); 9. Subjects vaccinated with a live vaccine within 30 days before the first administration, including, but not limited to, the following: mumps, rubella, measles, chickenpox/shingles (chickenpox), yellow fever, rabies, Bacille Calmette-Guerin (BCG) and typhoid vaccine (inactivated virus vaccine allowed); 10. Subjects who previously received PD-1/PD-L1 drug treatment or treatment of another drug targeting T cell receptors (such as CTLA-4 and OX-40); 11. Subjects who have had a severe allergic reaction to other monoclonal antibodies; 12. Subjects who have a history of severe allergies to pemetrexed, paclitaxel or albumin paclitaxel or docetaxel, cisplatin, carboplatin, recombinant human endostatin active ingredients, or preventive medications; 13. Subjects who are known to have serious or uncontrolled underlying diseases; 14. Subjects presenting malignant tumors other than NSCLC within 5 years before the first administration. Malignant tumors with negligible risk of metastasis or death (e.g., expected DFS> 5 years) and expected curative results after treatment (e.g., fully treated cervical carcinoma in situ, basal or squamous cell skin cancer, radical surgery treated ductal carcinoma in situ) can be excluded.

15. Subjects with grade III-IV congestive heart failure (New York Heart Association classification) and poorly controlled and clinically significant arrhythmia; 16. Subjects who have experienced any arterial thrombosis, embolism or ischemia, such as myocardial infarction, unstable angina, cerebrovascular accident, or transient ischemic attack, within 6 months before selection for treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 42 (Estimated)
Dates: Start 2022-05-15 (Estimated); Primary Completion 2023-05-15 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
MPR rate | 0-36months
  Major pathological reaction (MPR), defined as remaining viable tumor cells ≤ 10% at surgical resection of the primary tumor.MPR rate, defined as the proportion of intention-to-treat (ITT) population reaching MPR.

SECONDARY OUTCOMES:
the event-free survival (EFS) | 0-36months
  Event-free lifetime (EFS), defined as the time from the beginning of group entry to the occurrence of any of the following events
the complete pathological remission rate (pCR) | 0-36months
  pCR, defined as the absence of any surviving primary tumor cells on surgical removal of the primary tumor.
the disease-free survival (DFS) | 0-36months
  DFS, defined as the time from enrollment to local or distant recurrence (including the occurrence of new primary NSCLC) or death from any cause, whichever occurs first.
the 3-year survival rate and overall survival (OS) | 0-36months
  OS, defined as the time from treatment to the death of the subject due to any cause.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0, AEs, TEAEs, SAEs,irAEs | 0-36months
  The incidence and severity of all AEs, treatment-emergent AEs (TEAEs), serious AEs (SAEs), and immune-related AEs (irAEs), and their correlation with study drugs.

CONTACTS AND LOCATIONS:
Locations (1):
- the second Xiangya hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No